CLINICAL TRIAL: NCT02486939
Title: An Open-Label Safety Extension Study (OLSES) Evaluating the Long Term Safety and Durability of Response of CHS-0214 (CHS-0214-05)
Brief Title: A Long Term Safety Extension Study (CHS-0214-05)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHS-0214-05
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2017-11

CONDITIONS: Rheumatoid Arthritis; Plaque Psoriasis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CHS-0214 (Experimental): CHS-0214 50 mg weekly
  Interventions: Drug: CHS-0214

INTERVENTIONS:
Drug: CHS-0214 — Open label

SUMMARY:
An Open-label, Safety Extension Study (OLSES) evaluating the longer-term safety and durability of response of subjects who completed 48 weeks of evaluations in the confirmatory safety and efficacy studies, CHS 0214-02 or CHS-0214-04, evaluating CHS-0214 in patients with rheumatoid arthritis (RA) and plaque psoriasis (PsO), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Have completed 48 weeks of evaluations in CHS-0214-02 and, at Week 48, had at least an ACR20, or completed 48 weeks of evaluations in CHS-0214-04 and, at Week 48, had at least a PASI-50

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Finck, MD, Study Director — Coherus Oncology, Inc.
Locations (1):
- Oribe Clinic of Rheumatism and Medicine, Ōita, Oita Prefecture, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- CHS-0214-02 -RA: RA Participants
- CHS-0214-04 - PsO: PsO Participants
Period: Overall Study
Arm/Group | CHS-0214-02 -RA | CHS-0214-04 - PsO
Started | 225 | 134
Completed | 224 | 132
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- CHS-0214-02-RA: RA Participants
- CHS-0214-04-PsO: PsO Participants
- Total: Total of all reporting groups
Arm/Group | CHS-0214-02-RA | CHS-0214-04-PsO | Total
Number analyzed (Participants) | 224 | 132 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.28) | 45.9 (13.2) | 49.9 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 31 | 201
  Male | 54 | 101 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 222 | 128 | 350
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 167 | 9 | 176
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 108 | 158
  More than one race | 0 | 13 | 13
  Unknown or Not Reported | 7 | 2 | 9
Height [Mean (Standard Deviation); unit: Centimeters] | 162.1 (8.7) | 172.2 (10.71) | 165.9 (10.83)
Weight [Mean (Standard Deviation); unit: Kilograms] | 65.58 (17.604) | 92.19 (21.593) | 75.58 (23.599)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: "kg/m^2"] | 24.73 (5.287) | 31.06 (7.238) | 27.09 (6.823)

OUTCOME MEASURES:

1. Primary Outcome: Durability of Response (Maintenance of an ACR20 Response or Greater), Which Was Measured at Each Visit in Subjects of RA
Description: The ACR20 is a composite endpoint based on the following assessments: 66/68 swollen joint count (SJC) or tender joint count (TJC), Subject's pain assessment (SPA)-visual analog scale (VAS),Subject's global assessment of disease activity (SGA)-VAS,Physician's global assessment of disease activity (PGA)-VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI), and High sensitivity C-reactive protein (hs-CRP).The baseline value to assess the ACR20 during this study was the same baseline value used to assess the ACR20 during the parent study (ie, the Week 0 assessment in the parent study).
  Subjects were considered an ACR20 responder at a visit if compared to baseline in the parent study (CHS-0214-02) they achieved: At least 20% decrease in SJC, At least 20% decrease in TJC, and At least 20% improvement in at least 3 of the following 5 measures: C-reactive protein, HAQ-DI, SPA (using a VAS) for pain,SGA (using a VAS), orPGA (using a VAS).
Time Frame: 48 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CHS-0214-02 -RA
Number analyzed (Participants) | 224
Participants | 117

2. Primary Outcome: In Subjects With PsO, Durability of Response (Maintenance of PASI-50 Response or Greater), Which Was Measured at Each Visit.
Description: All PASI score assessors must have demonstrated proficiency at performing the PASI. Every attempt was made to use the same assessor for each subject throughout the study. n subjects with PsO, durability of response (maintenance of a PASI-50 response or greater at each assessment) was based on scoring the PsO lesions on a scale of 0 to 4 for 3 characteristics: erythema, induration, and desquamation, and within 4 anatomical regions: head, trunk, upper extremities, and lower extremities. Within each of these regions, the area of involvement was scored on a scale of 0 to 6, with the total score being a weighted average, and weights defined by the area of involvement. The clinician assessed the subject's PsO lesions according to the PASI and provided this score within the case report form at Weeks 0 (as the Week 48 assessment of the parent study), 4, 12, 24, 36, and 48. Subjects were classified as having a PASI-50 response based upon 50% reduction from baseline of the parent study.
Time Frame: Week 0,4,12,24,36,48
Measure: Count of Participants; unit: Participants
Arm/Group | CHS-0214-04 - PsO
Number analyzed (Participants) | 132
Participants | 94

3. Secondary Outcome: Disease Activity Score Using 28 Tender and Swollen Joint Counts, High Sensitivity C-reactive Protein, and Subject's Global Assessment of Disease Activity (DAS28-CRP[4]) <3.2 (ie, Low Disease Activity) at All Visits for All Subjects With RA.
Description: The DAS28-CRP(4) is a composite score (ranging from 0 to 9.4) calculated using the results of the TJC (using a 28 joint subset), SJC (using a 28 joint subset), hs-CRP level (mg/L), and SGA (0 to 100 scale). The DAS28-CRP(4) was calculated using the following formula:0.56*sqrt(28TJC) + 0.28*sqrt(28SJC) + 0.36*ln(CRP+1) + 0.014* SGA + 0.96. For DAS28-CRP(4), scores indicating high disease activity are >5.1; low disease activity are <3.2;and remission are <2.6.
Time Frame: 108 Weeks
Measure: Number; unit: participants
Arm/Group | CHS-0214-02 -RA
Number analyzed (Participants) | 224
participants
  Week 4 | 192
  Week 12 | 190
  Week 24 | 189
  Week 36 | 188
  Week 48 | 184
  Week 60 | 139
  Week 72 | 140
  Week 84 | 121
  Week 96 | 48
  Week 108 | 34
  Follow Up Visit | 5

4. Secondary Outcome: DAS28-CRP(4) <2.6 (ie, Remission) on All Visits After DAS28-CRP(4) <2.6 Was Achieved for Subjects With RA.
Description: as for outcome 3
Time Frame: 48 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CHS-0214-02 -RA
Number analyzed (Participants) | 224
Participants | 135

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting on Day 0 and collected at Day 28 (Week 4), Day 84 (Week 12), Day 168 (Week 24), Day 252 (Week 36), Day 336 (Week 48) and Day 364 or 28 days post last dose (Week 52 or 4 weeks post last dose) for subjects with rheumatoid arthritis and plaque psoriasis.
Description: Adverse events related to study drug injection sites were assessed at each visit and recorded by subjects in the eDiary following each injection through Week 48.
Arm/Group | CHS-0214-02-RA | CHS-0214-04-PsO
All-Cause Mortality (participants affected / at risk) | 1/224 | 0/132
Serious Adverse Events (participants affected / at risk) | 18/224 | 7/132
Other Adverse Events (participants affected / at risk) | 117/224 | 34/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHS-0214-02-RA (N=224) | CHS-0214-04-PsO (N=132)
Herpes Zoster (Infections and infestations) | 1 | 0 (0)
Pneumonia (Infections and infestations) | 2 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Temporal Lobe Epilepsy (Nervous system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 1
Arrythmia (Cardiac disorders) | 1 | 0
Spondylotlisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CHS-0214-02-RA (N=224) | CHS-0214-04-PsO (N=132)
Bronchitis (Infections and infestations) | 15 | 1
Influenza (Infections and infestations) | 15 | 9
Pharyngitis (Infections and infestations) | 13 | 2
Upper Respiratory Infection (Infections and infestations) | 21 | 16
Urinary Tract Infection (Infections and infestations) | 13 | 3
Stomatitis (Gastrointestinal disorders) | 14 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 0
Contusion (Injury, poisoning and procedural complications) | 12 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02486939/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT02486939/SAP_001.pdf